CLINICAL TRIAL: NCT05597501
Title: Manual-based Psychosocial Group Interventions for Coping With the Covid-19 Pandemic and Other Crises
Brief Title: Covid-Intervention-Study
Acronym: CIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department for Psychosomatic Medicine and Psychotherapy, University for Continuing Education Krems (Other)
Responsible Party: Principal Investigator, Carina Dinhof, Research assistant, Department for Psychosomatic Medicine and Psychotherapy, University for Continuing Education Krems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21/2021-2024
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Psychosocial Intervention
Keywords: manual-based group intervention; short-term intervention; covid-19; crisis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT (cognitiv behavioural-therapy)-based (Active Comparator): weekly psychosocial group-intervention (8 weeks) based on a CBT-manual
  Interventions: Behavioral: manual-based group interventions
- integrative therapy (Active Comparator): weekly psychosocial group-intervention (8 weeks) based on a integrative therapy manual
  Interventions: Behavioral: manual-based group interventions
- Existential Analysis and Logotherapy (Active Comparator): weekly psychosocial group-intervention (8 weeks) based on a Existential Analysis and Logotherapy manual
  Interventions: Behavioral: manual-based group interventions

INTERVENTIONS:
Behavioral: manual-based group interventions — weekly group interventions (90min) following manuals of either CBT, integrative therapy or existential analysis&logotherapy

SUMMARY:
The goal of this invention study is test and compare short-term manual-based psychosocial group interventions in die Austrian population suffering from stresses and strains due to the Covid-19 Pandemic and other crises.

The main question it aims to answer: Does short-term manual-based psychosocial group interventions improve the mental well-being of the participants?

Participants will attend weekly a manual-based group (8 weeks) and answer online-questionnaires and surveys (pseudonymized).

ELIGIBILITY:
Inclusion Criteria:

* above 18 years with psychosocial stresses and strains due to covid-19 pandemic and other crises

Exclusion Criteria:

* suicidal tendency
* insufficient knowledge of the German language
* psychotic episode
* no internet-access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Positive Mental Health Scale (PMH) | Screening - Start Intervention - after 8 weeks intervention - 4 months follow-up

SECONDARY OUTCOMES:
WHO-Five Well-Being Index (WHO-5) | Screening - Start Intervention - after 8 weeks intervention - 4 months follow-up
Patient Health Questionnaire-9 (PHQ-9) | Screening - Start Intervention - after 8 weeks intervention - 4 months follow-up
Generalized Anxiety Disorder Scale-7 (GAD-7) | Screening - Start Intervention - after 8 weeks intervention - 4 months follow-up
Somatic Symptome Scale-8 (SSS-8) | Screening - Start Intervention - after 8 weeks intervention - 4 months follow-up
Stress Coping Inventars (SCI) | Screening - Start Intervention - after 8 weeks intervention - 4 months follow-up
Pereived Stress Scale (PSS) | Screening - Start Intervention - after 8 weeks intervention - 4 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Probst, Univ.Prof.Dr, Principal Investigator — University of Continuing Education Krems; Carina Dinhof, MSc., Principal Investigator — University of Continuing Education Krems; Rafael Rabenstein, MBA, MSc., Principal Investigator — University of Continuing Education Krems
Locations (1):
- University of Continuing Education Krems, Krems, Austria

IPD SHARING:
Plan to Share IPD: No